CLINICAL TRIAL: NCT05738941
Title: Interventional Radiology Strategies in Management of Painful Bony Lesions
Brief Title: Interventional Radiology in Bony Lesions
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kero Wagdy, principle investigator, Assiut University
Other Study IDs: bone interventional radiology
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Bone Lesion
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: radiofrequency ablation — 17-G length-adjustable electrode (RITA RF Electrode;) a 200-W RF generator is going to be used,under CT fluoroscopic guidance. The type of the electrode and the length of the active tip will be selected according to the size, location, and shape of the tumor, as well as the operator preference.ablation will be performed with 100 W energy for 30 seconds. The number of electrodes placed, ablation time per electrode, total ablation time, and total energy delivered to targets, as well as the temperature of the lesions, will be recorded. For lesions less than 3 cm, surgery was performed with one electrode , and for lesions of 3 cm or more, two or more electrodes were used . The procedure may be followed by injection of bone cement through the same working cannula, and a long working time will be delivered (STABILIT, Merit Medical Systems, Inc.) for the optimal filling of the bone lesion
Procedure: angioembolization — Use a 4- or 5-French diagnostic catheter for the initial angiogram and either continue to use this catheter for embolization where the feeding vessel is large or add a standard 2.3- to 2.5-French microcatheter as a coaxial technique .
  - Injection of embolizing material in the feeding vessels using gel foam , PVA or histoacryl according to the nature of the bony lesion

SUMMARY:
To explore the capability of the interventional radiology techniques in management of the painful bony lesions .

DETAILED DESCRIPTION:
Bone tumors may present as incidental findings, with pain or loss of function, or as fractures [1].

Interventional Radiology (IR) has experienced an exponential growth in recent years. Technological advances of the last decades have made it possible to use new treatments on a larger scale, with good results in terms of safety and effectiveness[2] .

Today, IR represents a minimally invasive option of treatment for benign bony lesions (osteoid osteoma [OO], osteoblastoma, periosteal chondroma, etc.) and for palliation of metastases involving bone and soft-tissue sites beyond the liver and lung in an always-increasing number of cases [3][4].

The aim of minimally-invasive ablation treatment is addressing the biological pain due to the stretching and irritation of the periosteum secondary to tumor growth and due to osteoclast-mediated bone resorption with the release of neurostimulating cytokines. The purpose of cementoplasty is to treat the mechanical pain for the instability from pathologic microfractures [5] Radiofrequency ablation (RFA) and cementoplasty are safe, feasible, and promising clinical option for the management of painful bony tumors that are challenging for their morphology and location [6].

Also , there is a broad range of indications for transarterial embolization (TAE) in primary or metastatic bone tumors: to reduce operative haemorrhagic risks, to simplify or allow more definitive surgery, or in the context of pain palliation, fever, bleeding, or hypercalcemic and other rheological factors[1].

ELIGIBILITY:
Inclusion Criteria:

1. Painful primary bone tumors .
2. Bone secondaries not amenable to radiation therapy .
3. histopathologically radioresistant bony tumors.
4. Painful osteoporotic vertebral fractures.

Exclusion Criteria:

* 1- Contraindications to contrast media 2- Raised renal chemistry or chronic kidney disease . 3- Pregnant patients . 4- Abnormal coagulation profile . 5- Contraindications to anesthesia .

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients coming to Assiut university hospitals with painful bony lesions fulfilling the inclusion criteria and need intervention
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
pain management | visual analogue score will be evaluated before the procedure and at 1-week and 3-, 6-, and 12-month follow-up outpatient office visits
  quantification of the pain before and after treatment through VAS ( visual analogue scale ) score .
  it is a score from (0) to (10) . The minimum value (0) means no pain and highest value (10) means worst pain possible . Higher scores mean worse outcome .

SECONDARY OUTCOMES:
The Functional Mobility Scale (FMS) | preoperatively and 1 month after the treatment to assess the effect of treatment on level of mobility and ability to walk
  assess the effect of treatment on level of mobility and ability to walk. A 4-point FMS classification is used: 4, bedridden; 3, use of wheelchair; 2, limited painful ambulation; 1, normal ambulation.
Local tumor control | performed 6 months after the treatment
  the absence of viable tissue enhancing at imaging within the entire tumor treated

CONTACTS AND LOCATIONS:
Overall Officials: Ehab Mousa, MD, Principal Investigator — Assiut University

REFERENCES:
- [Background] Owen RJ. Embolization of musculoskeletal bone tumors. Semin Intervent Radiol. 2010 Jun;27(2):111-23. doi: 10.1055/s-0030-1253510. PMID 21629401
- [Background] Sgalambro F, Zugaro L, Bruno F, Palumbo P, Salducca N, Zoccali C, Barile A, Masciocchi C, Arrigoni F. Interventional Radiology in the Management of Metastases and Bone Tumors. J Clin Med. 2022 Jun 7;11(12):3265. doi: 10.3390/jcm11123265. PMID 35743336
- [Background] Barile A, Arrigoni F, Zugaro L, Zappia M, Cazzato RL, Garnon J, Ramamurthy N, Brunese L, Gangi A, Masciocchi C. Minimally invasive treatments of painful bone lesions: state of the art. Med Oncol. 2017 Apr;34(4):53. doi: 10.1007/s12032-017-0909-2. Epub 2017 Feb 24. PMID 28236103
- [Background] Rosenthal D, Callstrom MR. Critical review and state of the art in interventional oncology: benign and metastatic disease involving bone. Radiology. 2012 Mar;262(3):765-80. doi: 10.1148/radiol.11101384. PMID 22357881
- [Background] Rybak LD, Rosenthal DI, Wittig JC. Chondroblastoma: radiofrequency ablation--alternative to surgical resection in selected cases. Radiology. 2009 May;251(2):599-604. doi: 10.1148/radiol.2512080500. Epub 2009 Mar 20. PMID 19304917
- [Background] Pusceddu C, De Francesco D, Ballicu N, Santucci D, Marsico S, Venturini M, Fior D, Moramarco LP, Faiella E. Safety and Feasibility of Steerable Radiofrequency Ablation in Combination with Cementoplasty for the Treatment of Large Extraspinal Bone Metastases. Curr Oncol. 2022 Aug 20;29(8):5891-5900. doi: 10.3390/curroncol29080465. PMID 36005203
- [Background] Koo JS, Chung SH. The Efficacy of Radiofrequency Ablation for Bone Tumors Unsuitable for Radical Excision. Clin Orthop Surg. 2021 Jun;13(2):278-285. doi: 10.4055/cios19179. Epub 2021 May 18. PMID 34094020
- [Background] Wang B, Zhang K, Zhang X, Yang S, Hu M, Li P, Yang W, Fan J, Xing C, Yuan Q. Microwave ablation combined with cementoplasty under real-time temperature monitoring in the treatment of 82 patients with recurrent spinal metastases after radiotherapy. BMC Musculoskelet Disord. 2022 Nov 29;23(1):1025. doi: 10.1186/s12891-022-05999-y. PMID 36443787